CLINICAL TRIAL: NCT07244068
Title: Effect of Mat Pilates on Pain and Postural Alignment in School Going Children With Upper Crossed Syndrome.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/MUSFERAIQBAL
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Children, Only; Upper Crossed Syndrome
Keywords: Postural Alignment; Craniovertebral angle; Thoracic Kyphosis angle; Mat Pilates; Upper Crossed Syndrome
MeSH Terms: conditions — Oculocerebral hypopigmentation syndrome type Preus

STUDY DESIGN:
Intervention Model Description: This randomized control clinical Trial is to evaluate the effect of mat Pilates on postural alignment and pain levels in school-going children with Upper Crossed Syndrome. The study will focus on assessing changes in head, neck, and shoulder alignment, as well as any reduction in musculoskeletal discomfort following a structured Pilates intervention in children of age 8-16.This clinical Trial will be in two groups A) Intervention group B) Control Group. From a total of 28 Participants , 14 will be performing Mat pilates and routine Physical Therapy(Group A) while the other 14 will be performing just routine Physical Therapy exercises (Group B). Data Analysis will be done on Statistical Package for the Social Sciences (SPSS) version 26.00.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mat Pilates+ RPT (Active Comparator): Experimental Group will receive Mat Pilates exercises and Routine Physical Therapy (baseline treatment). Baseline treatment will include stretching, strengthening and corrective exercises. Session duration will be 30 minutes, 10 to 12 exercises in form of 10 steps will be carried out per session, with no more than three repetitions of each exercise.
  Interventions: Other: Mat Pilates and Routine Physical Therapy
- Routie Physical Therapy (RPT) (Active Comparator): Control Group will receive stretching, strengthening and postural correction exercises .Every exercise will be for 30 seconds on and 30 seconds off, 3 times per day, total time about 30 minutes.
  Interventions: Other: Routine Physical Therapy (RPT)

INTERVENTIONS:
Other: Mat Pilates and Routine Physical Therapy — Group A will receive Pilates exercises and Routine Physical Therapy (baseline treatment). Baseline treatment will include stretching, strengthening and corrective exercises. Session duration will be 30 minutes, 10 to 12 exercises in form of 10 steps will be carried out per session, with no more than three repetitions of each exercise. The following is a detailed description of each exercise to be utilized in both treatments, along with its starting and ending positions and number of repetitions(24).
  1. Corrected neck alignment while lying on the back on a mat (use pillows if needed)
  2. Arm circles (both directions) on the mat.
  3. Diamond press
  4. Diamond press and lateral arm movement to back extension.
  5. Arm slides 90°:
  6. Arm circles on a tiny barrel while lying on back.
  7. Chair expansion.
  8. Lying prone, stabilize the scapula and pump arms up and down with lower back support.
  9. Straps for chest expansion.
  10. Kneel plank on a Swiss ball.
  Arms: Mat Pilates+ RPT
Other: Routine Physical Therapy (RPT) — Group B will receive stretching, strengthening and postural correction exercises as follows: Exercises for postural correction, stretches, and strengthening for the pectoralis major, elevator scapulae, upper trapezius, serratus anterior, rhomboids, and deep neck flexors muscles. -Every exercise will be for 30 seconds on and 30 seconds off, 3 times per day, - Push-ups and head-neck retraction were also included, total time about 30 minutes.
  Arms: Routie Physical Therapy (RPT)

SUMMARY:
This randomized control clinical Trial is to evaluate the effect of mat Pilates on postural alignment and pain levels in school-going children with Upper Crossed Syndrome. The study will focus on assessing changes in head, neck, and shoulder alignment, as well as any reduction in musculoskeletal discomfort following a structured Pilates intervention in children of age 8-16.This clinical Trial will be in two groups A) Intervention group B) Control Group. From a total of 28 Participants , 14 will be performing Mat pilates and routine Physical Therapy(Group A) while the other 14 will be performing just routine Physical Therapy exercises (Group B). Data Analysis will be done on Statistical Package for the Social Sciences (SPSS) version 26.00.

DETAILED DESCRIPTION:
The current study will be randomized control trial, data will be collected from Physical Therapy department of Ittefaq Hospital, Lahore. The study will include 28 participants equally divided into two groups and randomly allocated. Inclusion criteria for the study will be UCS patients with age between 8 to 16yrs of either gender. Patients with any recent history of injury, severe systemic disorder and physical or sensory deficit will be excluded from the study.Group A (Experimental Group) will receive Pilates exercises and Routine Physical Therapy (baseline treatment). Baseline treatment will include stretching, strengthening and corrective exercises. Session duration will be 30 minutes, 10 to 12 exercises in form of 10 steps will be carried out per session, with no more than three repetitions of each exercise.Group B (Control Group) will receive stretching, strengthening and postural correction exercises as follows: Exercises for postural correction, stretches, and strengthening for the pectoralis major, elevator scapulae, upper trapezius, serratus anterior, rhomboids, and deep neck flexors muscles. -Every exercise will be for 30 seconds on and 30 seconds off, 3 times per day, - Push-ups and head-neck retraction were also included, total time about 30 minutes. Outcomes to be analyzed will be Craniovertebral angle and Thoracic Kyphosis angle and Pain. Data collection will be done before and after the intervention. Tools used for data collection will be kinovea software for Craniovertebral angle and Thoracic Kyphosis angle and Visual analouge scale (VAS) for pain. Data will be analyzed through SPSS version 26.00.

ELIGIBILITY:
Inclusion Criteria:

* School going children
* Children of the age 8-16.
* Children having Thoracic Kyphosis angle under 20° and over 40 °,and Craniovertebral angle under 48°

Exclusion Criteria:

* Children with systemic disorders.
* Children with recent history of injury.
* Physical or sensory defecit(16)

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 28 (Estimated)
Dates: Start 2025-10-28 (Actual); Primary Completion 2026-06-02 (Estimated); Study Completion 2026-06-16 (Estimated)

PRIMARY OUTCOMES:
Kinovea Software | 5 Minutes
  Kinovea is a free 2D motion analysis software that can be used to measure Craniovertebral angle, thoracic kyphosis angle and lumbar lordosis. This low-cost technology has been used in sports sciences, as well as in the clinical and research fields. One interesting tool is that it can measure an object (or person) passing in front of the camera, taking into account the perspective between the camera and the recorded object.
Visual Analouge Scale | 1 minute
  A visual analogue scale (VAS) is a measurement tool that uses a straight line to rate the intensity of subjective feelings, most commonly pain. The line is typically 10 cm long, with one end representing the lowest level (e.g., "no pain") and the other end representing the highest level (e.g., "worst pain imaginable"). A patient marks the line to indicate their current sensation, and the distance from the zero point is used as a score, often out of 10.

CONTACTS AND LOCATIONS:
Overall Officials: Musfera Iqbal, MS-PT, Principal Investigator — Riphah International University
Locations (1):
- Ittefaq Hospital (TRUST), Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shadi N, Khalaghi K, Seyedahmadi M. Comparing the effects of Pilates, corrective exercises, and Alexander's technique on upper cross syndrome among adolescent girls student (ages 13-16): a six-week study. BMC Sports Sci Med Rehabil. 2024 Jun 28;16(1):143. doi: 10.1186/s13102-024-00933-2. PMID 38943175